CLINICAL TRIAL: NCT03391349
Title: Quantification of Proteomes: L-plastin , Lipocalin and Adiponectin in Subgingival Tissue Samples of Generalized Severe Chronic Periodontitis Patients With and Without Type II Diabetes Mellitus
Brief Title: Quantification of Proteomes: L-plastin , Lipocalin and Adiponectin in Chronic Periodontitis and Diabetic Subjects
Status: Completed | Type: Observational
Sponsor: Meenakshi Ammal Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr.Jaideep Mahendra, Professor and PhD guide, Meenakshi Ammal Dental College and Hospital
Other Study IDs: MADC/IRB-IX/2016/151
Record Dates: First submitted 2017-12-21; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Periodontal Diseases
Keywords: proteomes, chronic periodontitis
MeSH Terms: conditions — Periodontal Diseases; Chronic Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: GROUP I: 35 generalized severe chronic periodontitis subjects without type II diabetes mellitus and systemically healthy.
- Group II: GROUP II: 35 generalized severe chronic periodontitis subjects diagnosed with type II diabetes mellitus.

SUMMARY:
The quantification of the proteomes : L-plastin, lipocalin and adiponectin was analysed in the subgingival tissue samples of generalized severe chronic periodontitis patients with and without diabetes mellitus.The demographic and the periodontal parameters were assessed and the correlated with the quantification of the proteins. The mRNA expression was analyzed with RT-PCR and the quantification of protein was done using ELISA.

DETAILED DESCRIPTION:
The quantification of the proteomes : L-plastin, lipocalin and adiponectin was analysed in the subgingival tissue samples of generalized severe chronic periodontitis patients with and without diabetes mellitus.A total of 70 subjects with generalized severe chronic periodontitis were selected and divided into two groups. Group I comprised of 35 subjects who were diagnosed with generalized severe chronic periodontitis without any systemic conditions. Group II comprised of generalized severe chronic periodontitis patients with type II diabetes mellitus. Demographic variables such as age, weight, height, BMI and income and the clinical parameters such as plaque index, bleeding on probing, probing pocket depth and clinical attachment level were recorded. Subgingival tissue samples were collected from both the groups from the periodontal surgical site. The collected samples were subjected to further molecular analysis for the mRNA expression of L-plastin, lipocalin and adiponectin using RT-PCR and for their protein quantification using ELISA.The elevated levels of mRNA expression and elevated quantification of L-plastin and Lipocalin proteins in the subgingival tissue samples of generalized severe chronic periodontitis subjects with diabetes denoted the localized involvement of these molecules in the pathogenesis of both periodontitis and type II diabetes mellitus. Since adiponectin was reduced in periodontitis patients with type II diabetes mellitus, it can be used as an anti-inflammatory and anti-diabetic biomarker for the early identification of patients at risk for diabetes mellitus and periodontitis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing to participate in the study.
2. Male patients within the age group 35 to 60 years.
3. Patients having ≥ 10 natural teeth.
4. No history of long term antibiotic use in the past 6 months and no history of diabetes mellitus.

For Group I:

• Generalized severe chronic periodontitis subjects (30% or more sites with clinical attachment loss (CAL) ≥ 5mm) without type II diabetes mellitus.

For Group II:

• Generalized severe chronic periodontitis subjects (30% or more sites with clinical attachment loss (CAL) ≥ 5mm) diagnosed with type II diabetes mellitus (HbA1C levels ≥7%) for the past 5 years and is under oral medication.

Exclusion Criteria:

1. Patients with systemic conditions, such as cardiovascular and respiratory diseases, HIV infection, immunosuppressive patients and patients under chemotherapy.
2. Smokers and other behavioral factors which may influence the study.
3. Patients who had undergone periodontal therapy within the previous 6 months.
4. Female patients (due to hormonal changes and pregnancy which may alter the oral flora).

   -

Ages: 35 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only male subjects were included in the study. females were excluded as hormonal changes may alter the oral flora.
Study Population: All male patients within the age group of 35-60 years. The subjects were from the South Indian population.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2017-07-22 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
mRNA expression of L-plastin,lipocalin and adiponection | 9 months
  mRNA expression of L-plastin,lipocalin and adiponectin using Real Time PCR

SECONDARY OUTCOMES:
Quantify the levels of L-plastin, lipocalin and adiponectin | 9 months
  Quantify levels of L-plastin, lipocalin and adiponectin using ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Jaideep Mahendra, MDS,PhD, Study Director — Meenakshi Ammal Dental College

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozturk VO, Emingil G, Osterwalder V, Bostanci N. The actin-bundling protein L-plastin: a novel local inflammatory marker associated with periodontitis. J Periodontal Res. 2015 Jun;50(3):337-46. doi: 10.1111/jre.12212. Epub 2014 Jul 12. PMID 25040533